CLINICAL TRIAL: NCT05869240
Title: A Phase I/II, Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BPB-101 in Patients With Advanced Malignant Solid Tumors.
Brief Title: BPB-101 in Subjects With Metastatic or Locally Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-61811
Record Dates: First submitted 2023-04-23; First posted 2023-05-22 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor
Keywords: BPB101; solid tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPB-101 (Experimental)
  Interventions: Drug: BPB-101

INTERVENTIONS:
Drug: BPB-101 — Subjects will receive an intravenous infusion of BPB-101 in a pre-set dose escalation until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the trial.

SUMMARY:
This is a multi-center, open-label, Phase I/II clinical study of BPB-101 as monotherapy in patients with advanced solid tumors to evaluate the safety, pharmacokinetic characteristics and antitumor activity of BPB-101.

DETAILED DESCRIPTION:
This trial consist of 3 parts: dose escalation(phase Ia), dose expansion(phase Ib) and clinical expansion(phase II) part. The current trial is composed of dose escalation with accelerated titration and "3 + 3" cohort design (phase Ia), for which 1 to 6 subjects will be enrolled at each dose level depending on the occurrence of dose limiting toxicities (DLT), followed by a consecutive parallel-group expansion in selected dose levels (phase Ib) and selected solid tumor indications (phase II). Participants enrolled in Phase 2 will receive the Recommend Phase 2 Dose (RP2D) of BPB-101 (determined by phase Ia dose escalation and phase Ib dose expansion) until confirmed progression, unacceptable toxicity, or any criterion for stopping the study drug or withdrawal from the trial occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the trial and sign an informed consent form.
2. Male or female subjects aged between 18 and 75 years.
3. Subjects with cytologically or histologically confirmed advanced solid tumor for which no standard therapy is available or standard therapy has failed in dose-escalation phase; In the dose-expansion phase, subjects enrollment included, but not limited to, with non-small-cell lung, esophageal, colorectal, endometrial, melanoma, bladder, and breast cancers (actual enrollment could be determined based on available data).
4. Life expectancy >= 12 weeks.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Participants enrolled in the dose-escalation phase (phase Ia) must have evaluable disease per RECIST 1.1. Participants enrolled in the dose expansion and clinical expansion phase (phase Ib and II) must have at least one measurable disease per RECIST 1.1.
7. Adequate hematologic and organ function at screening, as follows:

   1. Absolute neutrophil count (ANC)≥1.5×10^9/L, Platelets≥100×10^9/L, Hemoglobin≥9g/dL(90g/L)
   2. Serum total bilirubin ≤1.5×upper limit of normal (ULN), unless liver cancer or liver metastases are present, then values must be ≤2×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, unless liver cancer or liver metastases are present, then values must be ≤5×ULN
   3. Serum creatinine≤1.5×ULN OR creatinine clearance (CrCl)≥50ml/min (using the Cockcroft-Gault formula)
   4. International normalized ratio (INR) and prothrombin time ≤1.5×ULN; And activated partial thromboplastin time (aPTT) ≤1.5×ULN.
8. Female subjects with childbearing potential must have a negative serum pregnancy test at screening (within 7 days of first dose of study drug). Female subjects with childbearing potential and male subjects with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the trial starting with the screening visit through 6 months after the last dose of study drug is received.

Exclusion Criteria:

1. Known hypersensitivity to any component and excipients of the investigational drug, or previous severe allergic reaction to any macromolecular monoclonal antibody.
2. Received anti-PD-1 or PD-L1 antibodies within 3 months prior to screening. Previously received treatment targeting TGF-β, TGF-β receptors, or GARP.
3. Received other antitumor therapies, such as chemotherapy, biological therapy, endocrine therapy, etc., within 4 weeks before the first dose. Local palliative treatment (such as local surgery or radiotherapy) for isolated lesions can be received without affecting the efficacy evaluation. Enrollment is permitted in the following cases:

   * Oral pyrimidine or small molecule targeted therapy drugs are used more than 2 weeks or 5 half-lives of the drug (whichever is longer) before the first dose.
   * Nitrosourea or mitomycin C are used more than 6 weeks before the first dose.
4. Major surgery within 4 weeks before first dose of study drug.
5. Systemic therapy with immunosuppressive agents within 2 weeks prior to the first dose of study drug or during the study, except for corticosteroid nasal sprays, inhalers, or ≤10 mg/day systemic prednisone and equivalent medications.
6. Previous malignant disease (other than the target malignancy to be investigated in the trial) within the last 5 years.Except for malignancies that can be expected to heal after treatment (including but not limited to, adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, or carcinoma in situ of the breast duct treated with radical surgery).
7. Presence of symptomatic central nervous system metastases, meningeal metastases, or spinal cord compression due to metastases. Except for patients with brain metastases who have symptoms before the first dose, but whose disease is stable for ≥ 4 weeks after treatment.
8. Subjects with a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer; Those with a history of melena and hematemesis within 2 months before administration; Researchers believe that visceral bleeding may occur.
9. Patients with large and uncontrolled pleural effusions, pericardial effusions, or abdominal effusions requiring repeated drainage.
10. Has an active autoimmune disease requiring systemic treatment within 2 years prior to initial medication.
11. Cardiovascular diseases of clinical significance, including:

    a. Clinically uncontrolled hypertension;

    The following conditions occurred within 6 months before the first medication:
    1. Congestive heart failure (New York Heart Association Grade III or IV);
    2. Arrhythmias or conduction abnormalities that require medical treatment. Note: Subjects with drug-controlled atrial fibrillation/atrial flutter and pacemaker controlled arrhythmia can be enrolled;
    3. Severe/unstable angina, coronary/peripheral bypass graft, or myocardial infarction; (Note: Severe angina is Grade III or IV of the Canadian Cardiovascular Society)
    4. Cerebrovascular accident or transient ischemic attack, transient myocardial ischemia;
    5. Any other arterial thrombosis or embolic event.
12. Severe active infection within 2 weeks prior to initial administration, or systemic anti-infection therapy lasting more than 7 days after intravenous use within 1 week prior to initial administration.
13. Toxicity due to previous antitumor therapy has not returned to CTCAE 5.0 level ≤1 (except for toxicity such as alopecia where the investigator determined no safety-related risk).
14. There is active tuberculosis, or interstitial lung disease requiring treatment.
15. History of bone marrow allotransplantation or solid organ transplantation.
16. HIV-positive or active syphilis infection.
17. Have active hepatitis B and C.
18. Pregnant or lactating women.
19. Have received live or attenuated vaccine within 180 days prior to initial administration of study drug (Note: Inactivated virus vaccine is allowed. Seasonal flu vaccines that do not contain live viruses are allowed. Inactivated COVID-19 vaccine is allowed, but needs to be eluted for 1 week before first administration).
20. Any other disease or condition of clinical significance that the investigator believes may affect protocol compliance or the subject's signing of informed consent, or may be inappropriate for participation in the clinical trial.
21. Inability or unwillingness to follow the research and/or follow-up procedures outlined in the programme.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-08-02 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
DLT of BPB-101 | Up to 21 days after first treatment in Phase Ia
  DLT is defined as a dose-limiting toxicity event occurring during the DLT observation period that, as determined by the Investigator and/or Sponsor to be at least possibly related to BPB-101, is classified using NCI-CTCAE version 5.0 as conforming to adverse events (AEs) or laboratory anomalies specified in the protocol.
Maximum Tolerated Dose (MTD) of BPB-101 | Up to 21 days after first treatment in Phase Ia
  MTD was defined as the maximum dose of <1/3 DLT events observed in patients with evaluable DLT events (i.e., 1 in 6 patients at most).
RP2D of BPB-101 | Throughout Phase Ia and Ib，approximately 2 years
  RP2D is determined based on safety, tolerability, pharmacokinetics and efficacy data.
Number of subjects with adverse events (AEs) | Up to 30 days after last treatment
  An Adverse Event (AE) is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship.

SECONDARY OUTCOMES:
Dose Escalation and Expansion Part: Maximum concentration (Cmax) | Predose ,0, 2, 6, 24, 48, 168 and 336 hours post dose at cycle 1 and 3 (each cycle is 21 days); predose at cycle 2, 4 and every 4 cycles after cycle 8 until progression or end of the treatment whichever occur first, assessed up to 2 years.
  Serum BPB-101 concentrations measured throughout the study.
Dose Escalation and Expansion Part: Minimum concentration (Cmin) | Predose ,0, 2, 6, 24, 48, 168 and 336 hours post dose at cycle 1 and 3 (each cycle is 21 days); predose at cycle 2, 4 and every 4 cycles after cycle 8 until progression or end of the treatment whichever occur first, assessed up to 2 years.
  Serum BPB-101 concentrations measured throughout the study.
Dose Escalation and Expansion Part: Area under the concentration-time curve from zero to last sampling time (AUC0-t) | Predose ,0, 2, 6, 24, 48, 168 and 336 hours post dose at cycle 1 and 3 (each cycle is 21 days); predose at cycle 2, 4 and every 4 cycles after cycle 8 until progression or end of the treatment whichever occur first, assessed up to 2 years.
  Serum BPB-101 concentrations measured throughout the study.
Dose Escalation and Expansion Part: Half-life (T1/2) | Predose ,0, 2, 6, 24, 48, 168 and 336 hours post dose at cycle 1 and 3 (each cycle is 21 days); predose at cycle 2, 4 and every 4 cycles after cycle 8 until progression or end of the treatment whichever occur first, assessed up to 2 years.
  Serum BPB-101 concentrations measured throughout the study.
Immunogenicity of BPB-101 | Predose of cycle 1, 2, 3, 4 (each cycle is 21 days), and every 4 cycles after cycle 8 until progression or end of the treatment whichever occur first, assessed up to 2 years.
  Serum concentrations of anti-BPB 101 antibody measured throughout the study.
Objective Response Rate (ORR) | Evaluated throughout the protocol, for the duration of the trial, up to approximately 2 years
  Defined as the percentage of participants in the analysis population who had a Complete Response (CR) or Partial Response (PR) per iRECIST and RECIST 1.1(Phase 2 only).
Duration of Response (DOR) | Evaluated throughout the protocol, for the duration of the trial, up to approximately 2 years
  Defined as time from first observation of response to first observation of documented disease progression (or death) per iRECIST and RECIST 1.1(Phase 2 only)
Disease Control Rate (DCR) | Evaluated throughout the protocol, for the duration of the trial, up to approximately 2 years
  Defined as proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD) per iRECIST and RECIST 1.1(Phase 2 only)
Time to Response (TTR) | Evaluated throughout the protocol, for the duration of the trial, up to approximately 2 years
  Defined as the time from the first dose date to first observation of response per iRECIST and RECIST 1.1(Phase 2 only).
Progression-free Survival (PFS) | Evaluated throughout the protocol, for the duration of the trial, up to approximately 2 years
  Defined as time from first treatment administration to first observation of documented disease progression (or death）, per iRECIST and RECIST 1.1(Phase 2 only).
Overall survival (OS) | Evaluated throughout the protocol, for the duration of the trial, up to approximately 2 years
  Defined as time from start of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Study Chair — Sun Yat-sen University
Locations (4):
- China (4):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Sichuan Academy of Medical Sciences-Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No